CLINICAL TRIAL: NCT00417859
Title: Total Knee Arthroplasty: Comparison of Fixed and Mobile Bearings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Brigitte Jolles, MD, Prof, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HO 218/01
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- TKA mobile (Active Comparator): TKA mobile
  Interventions: Device: Total knee arthroplasty: mobile bearing
- TKA (No Intervention): TKA fix

INTERVENTIONS:
Device: Total knee arthroplasty: mobile bearing — Total knee arthroplasty: mobile bearing
  Arms: TKA mobile

SUMMARY:
The goal of this study is to provide gait parameters as a new objective method to assess total knee arthroplasty outcome between patients with fixed- and mobile-bearing, using an ambulatory device with minimal sensor configuration.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a primary unilateral knee osteoarthritis and requiring a knee replacement
* Informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2004-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Jolles, MD MSc, Principal Investigator — HOSR
Locations (1):
- HOSR, Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 patients were excluded
Groups:
- TKA Mobile: TKA mobile
  Total knee arthroplasty with mobile bearing implant.
- TKA Fix: Total knee arthroplasty with fixed bearing implant.
Period: Overall Study
Arm/Group | TKA Mobile | TKA Fix
Started | 26 | 30
Completed | 26 | 29
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TKA Fix: TKA fix
- Total: Total of all reporting groups
Arm/Group | TKA Mobile | TKA Fix | Total
Number analyzed (Participants) | 26 | 30 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.3) | 70.2 (7.1) | 68.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 9 | 18 | 27

OUTCOME MEASURES:

1. Primary Outcome: Gait Stride Length
Description: distance in meters of gait stride lenght measured by a data logger with five inertial sensors
Time Frame: 5years
Measure: Mean (Inter-Quartile Range); unit: meters
Groups:
- Preoperative: preoperative stride lenght of all participants
- 5 Years: stride lenght at 1 year following TKA of all participants
Arm/Group | Preoperative | 5 Years
Number analyzed (Participants) | 26 | 29
meters | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3]
Statistical Analysis 1: Comparison: Preoperative vs 5 Years; FB group was designated the control group. We determined a sample size based in clinical criteria. Using an α of 0.05 and β of 0.8, the required sample size was calculated to be 24 patients in each group to achieve a power of 80%. Descriptive analysis was completed on demographic information and clinical and radiological outcomes. Nonparametric tests (Wilcoxon's signed ranks or rank sum tests) were used for comparison of scores. The chi-squared test was used for dichotomous variables; Test type: Superiority; p = 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: EuroQoL Quality of Life Scale (EQ-5D)
Description: The EQ-5D is a measure of self-reported health outcomes that is applicable to a wide range of health conditions and treatments. It consists of two parts: a descriptive system (Part I) and a visual analogue scale (VAS) (Part II). Part I of the scale consists of 5 single-item dimensions including: mobility, self care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has a 3 point response scale designed to indicate the level of the problem. Part II uses a vertical graduated VAS (thermometer) to measure health status, ranging from worst imaginable health state to best imaginable health state. T.
  Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable). The score from Part II can be used to track changes in health, on an individual or group level, over time.
Time Frame: 5years
Population: data collected in 25 patients on each group (as this a patient reported outcome, thr data was missing in some of the cases)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TKA Mobile | TKA Fix
Number analyzed (Participants) | 25 | 25
score on a scale | 75.3 (17.5) | 79.9 (18.0)

3. Secondary Outcome: Semi-objective Evaluation Knee Sciety Score (KSS) Clinical Outcome Measures
Description: Scoring system to clinically rate the knee abefore and after TK, scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Time Frame: 5years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TKA Mobile | TKA Fix
Number analyzed (Participants) | 25 | 25
score on a scale | 51.7 (12.8) | 49.3 (19.4)

4. Secondary Outcome: Number of Participants With Dislocation
Description: count of numbers of dislocated implants.
Time Frame: 5years
Measure: Count of Participants; unit: Participants
Arm/Group | TKA Mobile | TKA Fix
Number analyzed (Participants) | 26 | 29
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | TKA Mobile | TKA Fix
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TKA Mobile (N=25) | TKA Fix (N=25)
postoperative varus knee laxity due to a deficiency in the fibular collateral ligament (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No